CLINICAL TRIAL: NCT01180465
Title: A Multi-center, Randomized, Double-masked, Placebo-controlled, Dose-ranging, Study of the Safety and Efficacy of Subcutaneous Injections of LIPO-102 Compared With Placebo for the Reduction of Abdominal Subcutaneous Adiposity
Brief Title: A Dose-ranging, Study of the Safety and Efficacy of Subcutaneous Injections of LIPO-102 Compared With Placebo for the Reduction of Abdominal Subcutaneous Adiposity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neothetics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LIPO-102-CL-09; LIPO-102-CL-09
Record Dates: First submitted 2010-08-10; First posted 2010-08-12 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Weight
Keywords: Treatment of abdominal adiposity
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- LIPO-102 High (Experimental)
  Interventions: Drug: LIPO-102
- LIPO-102, Low (Experimental)
  Interventions: Drug: LIPO-102 Low
- LIPO-102; Placebo (Placebo Comparator)
  Interventions: Drug: LIPO-102, Placebo

INTERVENTIONS:
Drug: LIPO-102 — LIPO-102 High dose
  Arms: LIPO-102 High
Drug: LIPO-102 Low — LIPO-102 Low dose
  Arms: LIPO-102, Low
Drug: LIPO-102, Placebo — Placebo
  Arms: LIPO-102; Placebo

SUMMARY:
LIPO-102 is under evaluation for treatment of abdominal adiposity

ELIGIBILITY:
Inclusion Criteria:

* 18 - 50 years old inclusive
* Localized area of abdominal subcutaneous adiposity of Grade 3 or above on the P-PNS or C-PNS
* BMI < 25kg/m sq
* Stable diet and exercise and body weight

Exclusion Criteria:

* Prior treatment of abdominal subcutaneous adipose tissue
* Females within 12 months postpardum
* Known hypersensitivity to the drugs or components

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2010-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Safety | 8 weeks treatment and 1 week follow up
  physical exam, ECG, vital signs, clinical assessment is injection site, clinical laboratory tests, and adverse events
Change in abdominal circumference | 8 weeks
  abdominal circumference

SECONDARY OUTCOMES:
photographic assessment | 8 weeks
  abdominal circumference and volume reduction assessment
Abdominal subcutaneous adiposity questionnaire | 8 weeks
  Patient reported outcome
Patient and clinician photo numeric scale | 8 weeks
  patient and physician reports of change
Patient global assessment of severity scale | 8 weeks
  patient reports of change in severity

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - San Diego, California
  - New York, New York